CLINICAL TRIAL: NCT04116658
Title: A Multicenter, Open-Label, First-in-Human, Phase 1b/2a Trial of EO2401, a Novel Multipeptide Therapeutic Vaccine, With and Without Check Point Inhibitor, Following Standard Treatment in Patients With Progressive Glioblastoma
Brief Title: First-in-Human, Phase 1b/2a Trial of a Multipeptide Therapeutic Vaccine in Patients With Progressive Glioblastoma
Acronym: ROSALIE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Enterome (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EOGBM1-18
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma, Adult
Keywords: Glioblastoma; Vaccine; Nivolumab; Bevacizumab; Safety; Tolerability
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Multiple dose of EO2041 monotherapy followed by continued EO2401 in combination with nivolumab
  Interventions: Biological: Multiple dose of EO2401
- Cohort 2 (Experimental): Multiple dose of EO2041 in combination with nivolumab
  Interventions: Biological: Multiple dose of EO2401
- Cohort 3 (Experimental): Multiple dose of EO2041 in combination with nivolumab and bevacizumab
  Interventions: Biological: Multiple dose of EO2401

INTERVENTIONS:
Biological: Multiple dose of EO2401 — Multiple dose administration of EO2401 coadministered with or without nivolumab (and bevacizumab, US only) during the priming phase

SUMMARY:
The purpose of this study is to assess the safety, tolerability, immunogenicity, and preliminary efficacy of EO2401 in patients with unequivocal evidence of progressive or first recurrent glioblastoma.

DETAILED DESCRIPTION:
This is a multicenter, Phase 1b/2a, First-In-Human study to assess the safety, tolerability, immunogenicity, and preliminary efficacy of EO2401 in patients with unequivocal evidence of progressive or first recurrent glioblastoma.

EO2401 is an innovative cancer peptide therapeutic vaccine based on the homologies between Tumor Associated Antigens and microbiome-derived peptides that will be administered alone and in combination with nivolumab, and nivolumab/bevacizumab to generate preliminary safety and efficacy data in patients with progressive glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unequivocal documented (including histological confirmation of Glioblastoma-GB- at the primary diagnosis) evidence of first progression/recurrence of GB on MRI, as defined by RANO criteria
2. Patients with :

   * for Cohorts 1, 2a, and 3: at least 1 measurable lesion
   * for Cohort 2b: no measurable enhancing disease
   * for Cohort 2c: documented recurrence of GB deemed to be candidate for surgery
3. Patients with an age ≥ 18 years old
4. Patients who are human leukocyte antigen (HLA)-A2 positive
5. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 or Karnofsky performance status ≥ 70
6. Patients should have received standard primary therapy, including surgery (biopsy, incomplete or complete resection), radiation, temozolomide, if applicable

   1. Radiation therapy must have been finished 28 days before first study treatment administration
   2. Patients who received temozolomide as adjuvant therapy must have stopped the treatment and have a wash-out period of 28 days before first study treatment administration (6 weeks for nitrosoureas and 5 half lives for experimental therapies)
   3. Patients with unmethylated methylguanine-DNA-methyltransferase (MGMT) promoter can be included even if they have not received temozolomide prior to the inclusion in this clinical study)
7. Female patients of childbearing potential must have a negative serum pregnancy test within 72 hours prior to dosing
8. Considering the embryofetal toxicity of the nivolumab shown on animals' models, the following recommendations for contraception must be followed:

   a. If not surgically sterile, female patients of childbearing potential age must use highly effective contraception from signing the Informed Consent Form (ICF) through 6 months after the last treatment dose administered. Highly effective contraception included: i. Combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation: Oral Intravaginal Transdermal ii. Progestogen-only hormonal contraception associated with inhibition of ovulation: Oral Injectable Implantable iii. Intrauterine device iv. Intrauterine hormone-releasing system v. Bilateral tubal occlusion vi. Sexual abstinence. In each case of delayed menstrual period (over 1 month between menstruations), confirmation of absence of pregnancy is strongly recommended. This recommendation also applies to women of childbearing potential with infrequent or irregular menstrual cycles.

   b. If not surgically sterile, male with female partner of childbearing potential must use condom from signing the ICF through 8 months after the last treatment dose administered. Males must ensure that their partners of childbearing potential use highly effective contraception also.
9. Patients having received the information sheet and who have provided written informed consent prior to any study-related procedures
10. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.

Exclusion Criteria:

1. Patients treated with dexamethasone > 2 mg/day or equivalent (i.e., 13 mg/day of prednisone) within 14 days before the first EO2401 administration, unless required to treat an adverse event (AE) Note: The criterion implios the patient should not receive treatment with dexamethasone > 2 mg/day or equivalent at the actual time of a screening visit (single time point assessment), and within 14 days before the first EO2401 administration (unless required to treat AE); the latter part of the criterion should be checked at the time of treatment start.
2. 2. Patients treated with radiotherapy, and cytoreductive therapy within 28 days (6 weeks for nitrosoureas) before the first EO2401 administration. In addition, patients should not have received any prior treatment with compounds targeting PD-1, PD-L1, CTLA-4, or similar compounds where general resistance against therapeutic vaccination approaches might have developed; also, patients should not have received systemic anti-tumor treatment or radiotherapy for their progressive or first recurrent GB.
3. Patients with tumors primarily located in the infra-tentorial segment
4. Patients with known radiological evidence of extracranial metastases
5. Patients with presence of new hemorrhage (excluding, stable Grade 1) or uncontrolled seizure
6. Patients with significant leptomeningeal disease
7. Patients with abnormal (≥ Grade 2 National Cancer Institute-Common Terminology Criteria for AEs [NCI-CTCAE] version 5.0) laboratory values for hematology, liver, and renal function (serum creatinine). In detail, the following values apply as exclusion criteria:

   1. Hemoglobin < 10 g/dL (6.2 mmol/L)
   2. White blood cell count decrease (< 3.0 × 109/L) or increase (> 10.0 × 109/L)
   3. Absolute neutrophil count decrease (< 1.5 × 109/L)
   4. Platelet count decrease (< 75 × 109/L)
   5. Bilirubin > 1.5 × upper limit of normal per local laboratory levels; note, patients with hypothyroidism only requiring hormone replacement therapy are permitted to enroll, also patients with abnormal laboratory values judged by the treating physician as clinically non-relevant.
   6. Alanine aminotransferase > 3 × ULN
   7. Aspartate aminotransferase > 3 × ULN
   8. Serum creatinine increase (> 1.5 × ULN)
   9. Abnormal thyroid function
8. For patients who are planned to receive bevacizumab:

   1. Patients with nephrotic syndrome
   2. Patients with proteinuria ≥ 2g/24 hours
   3. Patients with history or active gastrointestinal perforation and fistula
   4. Significant surgical procedure in the 4 weeks preceding the start of treatment or planned surgery
   5. Unhealed wound
   6. Patient with recent (4 weeks) history of hemoptysis of ½ teaspoon or more of red blood
   7. Thrombotic episode within 6 months
   8. Uncontrolled diabetes mellitus or hypertension
   9. Posterior reversible encephalopathy syndrome
9. Patients with persistent Grade 3 or 4 toxicities (according to NCI-CTCAE v5.0). Toxicities must be resolved since at least 2 weeks to Grade 1 or less. However, alopecia or other persisting toxicities Grade ≤ 2 not constituting a safety risk based on Investigator's judgment is acceptable
10. Patients with contraindication to contrast-enhanced MRI
11. Other malignancy or prior malignancy with a disease-free interval of less than 3 years except those treated with surgical intervention and an expected low likelihood of recurrence such as basal cell or squamous cell skin cancer, or carcinoma in situ. Patients with adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ are eligible
12. 12. Patients with clinically significant active infection, cardiac disease, significant medical or psychiatric disease/condition that, in the opinion of the Investigator, would interfere with the evaluation of EO2401 or interpretation of patient safety or study results or that would prohibit the understanding or rendering of informed consent (i.e. only consent able patients can be enrolled in the study) and compliance with the requirements of the protocol - including (but not limited to):

    1. Bacterial sepsis or other similarly severe infections
    2. New York Heart Association > Grade 2 congestive heart failure within 6 months prior to study entry
    3. Uncontrolled or significant cardiovascular disease, including:

    i. Myocardial infarction within 6 months prior to obtaining informed consent ii. Uncontrolled/unstable angina within 6 months prior to obtaining informed consent iii. Diagnosed or suspected congenital long QT syndrome iv. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) d. Stroke within 6 months prior obtaining informed consent e. Concurrent neurodegenerative disease f. Dementia or significantly altered mental status.
13. Patients with suspected autoimmune or active autoimmune disorder or known history of an autoimmune neurologic condition (e.g., Guillain-Barré syndrome) Note, patients with vitiligo, type I diabetes mellitus, hypothyroidism due to autoimmune condition only requiring hormone replacement therapy, psoriasis not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
14. Patients with history of solid organ transplantation or hematopoietic stem cell transplantation
15. Patients with history or known presence of tuberculosis
16. Pregnant and breastfeeding patients
17. Patients with history or presence of human immunodeficiency virus and/or potentially active hepatitis B virus/hepatitis C virus
18. Patients who have received live or attenuated vaccine therapy used for prevention of infectious diseases including seasonal (influenza) vaccinations within 4 weeks of the first dose of study drug
19. Patients with a history of hypersensitivity to any excipient present in the pharmaceutical form of investigational medicinal product
20. Patients under treatment with immunostimulatory or immunosuppressive medications, including herbal remedies, or herbal remedies known to potentially interfere with major organ function
21. Patients with known drug and alcohol abuse
22. Patients with known or underlying medical or psychiatric condition that, in the Investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or AEs
23. Patients who have received treatment with any other investigational agent, or participation in another clinical trial (clinical trial including active interventions are prohibited; participation in clinical trials for data collection purposes only are permitted) within 28 days prior to first study treatment administration and during the treatment period. Note, for investigational agents there should be a wash-out period of at least 28 days, or 5 half-lives if longer, before first study treatment administration
24. Patients deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Paillarse, Study Director — Enterome
Locations (10):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States
- France (2):
  - Centre Georges François Leclerc, Dijon
  - Hôpital Pitié-Salpétrière, Paris
- Germany (5):
  - Klinik und Poliklinik für Neurologie Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Frankfurt Goethe-Universität Dr. Senckenbergisches Institut für Neuroonkologie, Frankfurt am Main
  - Neurologische Klinik & Nationales Zentrum für Tumorenerkrankungen Heidelberg Universitätsklinikum Heidelberg, Heidelberg
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Zentrum für Neuroonkologie Universitätsklinikum Tübingen, Tübingen
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institit Catala D'Oncologia - Hospital Duran i Reynals, L'Hospitalet de Llobregat

IPD SHARING:
Plan to Share IPD: Yes
Safety and survival data
Supporting Information: Study Protocol, SAP
Time Frame: Sep 2025
Access Criteria: Primary and key secondary outcome measures

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: EO2041 (1,2 mg) monotherapy followed by continued EO2401 in combination with nivolumab
- Cohort 2: EO2041 (1,2mg) in combination with nivolumab
- Cohort 3: EO2041 (1,2mg) in combination with nivolumab and bevacizumab
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 21 | 53 | 26
Completed | 21 | 53 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: EO2041 monotherapy followed by continued EO2401 in combination with nivolumab
- Cohort 2: EO2041 in combination with nivolumab
- Cohort 3: EO2041 in combination with nivolumab and bevacizumab
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 21 | 53 | 26 | 100
Age, Continuous [Median (Full Range); unit: years] | 58 [19 to 73] | 57 [18 to 78] | 60.5 [24 to 73] | 58 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 21 | 10 | 38
  Male | 14 | 32 | 16 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 19 | 46 | 24 | 89
  Unknown or Not Reported | 2 | 5 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 4 | 0 | 4
  White | 19 | 48 | 25 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of EO2401 Monotherapy, EO2401 in Combination With Nivolumab , EO2401 in Combination With Nivolumab and Bevacizumab
Description: Incidences of treatment-emergent Serious Adverse Events ( SAEs) using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0.
Time Frame: From treatment start up to study end, assessed up to 27.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 53 | 26
Participants | 9 | 8 | 8

2. Primary Outcome: Safety and Tolerability of EO2401 Monotherapy, EO2401 in Combination With Nivolumab , EO2401 in Combination With Nivolumab and Bevacizumab
Description: Incidences of treatment-emergent AEs (TEAEs) using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0.
Time Frame: From treatment start up to study end, assessed up to 27.5 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: EO2401 in combination with nivolumab
- Cohort 3: EO2401 in combination with nivolumab and bevacizumab
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 53 | 26
Participants | 21 | 51 | 26

3. Primary Outcome: Safety and Tolerability of EO2401 Monotherapy, EO2401 in Combination With Nivolumab , EO2401 in Combination With Nivolumab and Bevacizumab
Description: Incidences of deaths
Time Frame: From treatment start up to study end, assessed up to 44 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3: EO2401 in combination with nivolumab with bevacizumab
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 53 | 26
Participants | 20 | 46 | 23

4. Secondary Outcome: Evaluation of Survival
Description: Overall survival, defined as the time interval from the date of first study treatment administration to the date of death due to any cause
Time Frame: From treatment start up to study end, assessed up to 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 21 | 53 | 26
months | 9.6 [5.9 to 10.8] | 11.3 [9.0 to 13.7] | 12.1 [8.0 to 14.8]

5. Secondary Outcome: Assessment of the Immunogenicity of EO2316, EO2317, EO2318 (Three Components of the Therapeutic Vaccine), and Universal Cancer Peptide That Compose EO2401
Description: At least one positive response (proof of CD8 T cells specific for the EO2401 mimic peptides and/or for the tumor associated antigen (TAA) target peptides) in either of the used immunomonitoring assays (i.e. CD8 T cell expansion in peripheral blood measured by tetramers/flow cytometry, and Spot-Forming Cells by IFN-γ ELISPOT, both methods applied ex vivo, i.e. without prolonged in vitro stimulation and after in vitro stimulation)
Time Frame: 6 weeks after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 18 | 30 | 22
Participants | 17 | 29 | 20

ADVERSE EVENTS:
Time Frame: 44 months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 20/21 | 46/53 | 23/26
Serious Adverse Events (participants affected / at risk) | 9/21 | 8/53 | 8/26
Other Adverse Events (participants affected / at risk) | 20/21 | 51/53 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=21) | Cohort 2 (N=53) | Cohort 3 (N=26)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=21) | Cohort 2 (N=53) | Cohort 3 (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (6) | 4 (5)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 6 (9)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 3 (3) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (3) | 3 (3) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye haematoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Anal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (5)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (7) | 4 (6)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5) | 1 (1)
Asthenia (General disorders) | 2 (3) | 6 (13) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 15 (19) | 8 (9)
Gait disturbance (General disorders) | 0 (0) | 2 (3) | 5 (7)
General physical health deterioration (General disorders) | 4 (4) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 3 (4) | 0 (0)
Injection site discharge (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (2) | 5 (10) | 1 (1)
Injection site granuloma (General disorders) | 3 (3) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 1 (2) | 2 (2) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 6 (8) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (5) | 2 (2)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 5 (9) | 10 (25) | 13 (32)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Local reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical device site fistula (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (2) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 6 (10) | 5 (6)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (3) | 1 (1)
Acne pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 4 (6) | 6 (9)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 7 (8) | 7 (12)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 4 (4) | 8 (11)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 3 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (3) | 2 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 6 (6)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 5 (6) | 3 (3) | 3 (9)
Lymphocyte count decreased (Investigations) | 2 (6) | 7 (17) | 10 (29)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (5) | 4 (6)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 5 (8)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Thyroxine decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Thyroxine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 3 (5) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 6 (10)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 4 (10)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (8)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 3 (3)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alexia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 3 (5) | 9 (14) | 4 (4)
Apraxia (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Clumsiness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 4 (7) | 5 (5)
Dysdiadochokinesis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fine motor skill dysfunction (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 18 (32) | 9 (14)
Hemianopia (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Hemihypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 6 (7) | 6 (7) | 5 (10)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Language disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Monoparesis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 5 (5) | 3 (5)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 2 (6)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Quadrantanopia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (3) | 3 (4) | 7 (19)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Vibratory sense increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4) | 2 (2)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 2 (6) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 1 (3) | 4 (6)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 4 (4)
Learning disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mutism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 6 (13)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 5 (6)
Hypotension (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04116658/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT04116658/SAP_001.pdf